CLINICAL TRIAL: NCT02528877
Title: A Phase I Trial of Ruxolitinib Combined With Tacrolimus and Sirolimus as Acute Graft-versus-Host Disease (aGVHD) Prophylaxis During Reduced Intensity Allogeneic Hematopoietic Cell Transplantation in Patients With Myelofibrosis
Brief Title: Ruxolitinib Phosphate, Tacrolimus and Sirolimus in Preventing Acute Graft-versus-Host Disease During Reduced Intensity Donor Hematopoietic Cell Transplant in Patients With Myelofibrosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study design was revised so a new protocol will be opened.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14129; NCI-2015-01333 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14129 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Acute Myeloid Leukemia in Remission; Primary Myelofibrosis; Primary Myelofibrosis, Prefibrotic Stage; Secondary Acute Myeloid Leukemia; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fludarabine phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation; ruxolitinib; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (ruxolitinib phosphate, tacrolimus, sirolimus) (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV on days -9 to -5 and melphalan IV over 20 minutes on day -4. Beginning greater than 48 hours after completion of melphalan, patients undergo peripheral blood stem cell or bone marrow transplant according to standard guidelines on day 0.
  GVHD PROPHYLAXIS: Patients receive ruxolitinib phosphate PO BID on days -3 to 30 tapered to day 60, tacrolimus IV continuously or PO BID on days -3 to 100 , and sirolimus PO QD on day -3 to 100. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Drug: Ruxolitinib Phosphate; Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic bone marrow transplant
  Other Names: Allo BMT; Allogeneic BMT
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoeitic stem cell transplant
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo hematopoietic stem cell transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; RAPAMYCIN; SILA 9268A; WY-090217
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Prograf; Protopic

SUMMARY:
This phase I trial studies the side effects and best dose of ruxolitinib phosphate when given together with tacrolimus and sirolimus in preventing acute graft-versus-host disease during reduced intensity donor hematopoietic cell transplant in patients with myelofibrosis. Sometimes transplanted cells from a donor can attack the normal tissue of the transplant patient called graft-versus-host disease. Ruxolitinib phosphate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It may also reduce graft-versus-host disease by reducing inflammation and immune modulation. Giving ruxolitinib phosphate together with tacrolimus and sirolimus after transplant may prevent graft-versus-host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Among the dose levels tested, to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of ruxolitinib (ruxolitinib phosphate), when given in combination with tacrolimus and sirolimus (TAC/SIR) as acute graft-versus-host disease (aGVHD) prophylaxis as part of reduced intensity allogeneic hematopoietic cell transplant (HCT), in patients with myelofibrosis or other related myeloid neoplasm with marrow fibrosis.

SECONDARY OBJECTIVES:

I. To determine if the addition of ruxolitinib, to the standard aGVHD prophylactic regimen of TAC/SIR, is safe by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

II. To estimate the cumulative incidence of aGVHD and non-relapse mortality (NRM) at 100-days post transplant.

III. To estimate the cumulative incidence of chronic GVHD at 1- and 2-years post transplant.

IV. To characterize and evaluate hematologic recovery, donor cell engraftment and immune reconstitution by cell count and flow cytometry of lymphocyte subsets.

V. To estimate the probabilities of overall and progression-free survival (OS/PFS) at 1- and 2-years post transplant.

VI. To characterize changes in aGVHD biomarkers (regenerating islet-derived 3-alpha [Reg-3alpha], soluble tumor necrosis factor receptor I [sTNF RI], interleukin 2 receptor alpha [IL2Ralpha]), Janus-associated kinase (JAK)-regulated pro-inflammatory cytokines (i.e. interleukin [IL]-6, tumor necrosis factor [TNF] alpha, C-reactive protein [CRP], beta 2 microglobulin) and signal transducer and activator of transcription 3 (STAT3) phosphorylation (downstream of JAK signaling) over time and by aGVHD status/grade.

OUTLINE: This is a dose-escalation study of ruxolitinib phosphate.

PREPARATIVE REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -9 to -5 and melphalan IV over 20 minutes on day -4. Beginning greater than 48 hours after completion of melphalan, patients undergo peripheral blood stem cell or bone marrow transplant according to standard guidelines on day 0.

GVHD PROPHYLAXIS: Patients receive ruxolitinib phosphate orally (PO) twice daily (BID) on days -3 to 30 tapered to day 60, tacrolimus IV continuously or PO BID on days -3 to 100 , and sirolimus PO once daily (QD) on day -3 to 100. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary myelofibrosis intermediate or high risk by Dynamic International Prognostic Scoring System 26 (DIPSS26) in chronic or accelerated phase
* Transformed acute myeloid leukemia (AML) with marrow fibrosis is allowed, if AML is in complete remission after induction therapy
* Patients with a performance status of >= 70% on the Karnofsky scale
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for 1 year following transplant as per City of Hope standard operating procedure, (SOP) for allogeneic transplantation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Bone marrow and peripheral blood studies must be available for confirmation of diagnosis; cytogenetics, flow cytometry, and molecular studies (such as JAK-2, myeloproliferative leukemia [MPL] and calreticulin [CALR] mutational status) will be obtained as per standard practice
* Bone marrow aspirates/biopsies should be performed within 23 ± 7 days from registration to confirm disease remission status
* All candidates for this study must have a human leukocyte antigen (HLA) (A, B, C, DR) identical siblings who is willing to donate bone marrow or primed blood stem cells or an 8/8 allele-matched unrelated donor
* All ABO blood group combinations of the donor/recipient are acceptable since even major ABO compatibilities can be dealt with by various techniques (red cell exchange or plasma exchange)
* A cardiac evaluation with an electrocardiogram showing no ischemic changes or abnormal rhythm and an ejection fraction of 50% established by multi gated acquisition scan (MUGA) or echocardiogram
* Patients must have creatinine of less than or equal to 1.5 mg/dL or creatinine clearance > 60 ml/min
* A bilirubin of up to 2.0 mg/dL, excluding patients with Gilbert's disease
* Patients should also have a serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) less than 5 times the upper limit of normal
* Pulmonary function test including diffusing capacity of the lung for carbon monoxide (DLCO) will be performed; forced expiratory volume in 1 second (FEV1) and DLCO should be greater than 50% of predicted normal value
* All subjects must have the ability to understand and the willingness to sign a written informed consent that has been approved by the City of Hope (COH) Institutional Review Board (IRB); the patient, a family member and transplant staff physician (physician, nurse, and social worker) will meet at least once prior to the subject signing consent; during this meeting all pertinent information with respect to risks and benefits to donor and recipient will be presented; alternative treatment modalities will be discussed; the risks are explained in detail in the enclosed consent form
* Prior therapy with hydroxyurea, interferon, anagrelide, ruxolitinib, hypomethylating agents, Revlimid, thalidomide, steroids, other JAK inhibitors is allowed for AML patients who are back in chronic phase MPN, prior induction chemotherapy is allowed
* DONOR: Donor evaluation and eligibility will be assessed as per current City of Hope SOP

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ruxolitinib
* Patients with active 2nd malignancies other than myelofibrosis, AML, excised skin cancer, early stage cervical and prostate cancer
* Previous allogeneic hematopoietic stem cell transplantation
* Any psychiatric, social or compliance issues that, in the treating physician opinion, will interfere with completion of the transplant treatment and follow up
* Patients who have been treated with chemotherapy or radiation within two weeks of planned study enrollment; this does not include hydroxyurea or ruxolitinib, which may be continued until start of conditioning therapy
* Non-compliance defined as any subject, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events recorded using the modified Bearman scale and NCI CTCAE version 4.03 | Up to 2 years
  Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
MTD based on dose limiting toxicity recorded using the modified Bearman scale and National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 60 days post stem cell infusion
Recommended phase II dose of ruxolitinib phosphate, when given in combination with tacrolimus and sirolimus | Up to 60 days post stem cell infusion

SECONDARY OUTCOMES:
aGVHD graded and staged according to the Consensus grading | Up to 100 days post transplant
  The first day of acute GVHD onset at a certain grade will be used to calculate the cumulative incidence (grades II-IV). Calculated using the Gray method with prior death or relapse considered competing events.
Changes in expression levels of biomarkers | Baseline to up to day 100
  For all cytokines/biomarkers that are measured repeatedly over time, a nonparametric smoothing plot will be produced in the first step to view changes in the trend. Expression level changes on the onset of aGVHD from baseline measures will be correlated with aGVHD grade (0-1 vs 2-4 or 0-2 vs 3-4). Furthermore, GVHD biomarkers, Reg-3a, TNF R1, and a composite biomarker panel of 4 proteins (IL-2Ra, TNFR1, IL-8, and hepatocyte growth factor) will be correlated with survival outcomes in a continuous manner or dichotomized manner.
Chronic graft versus host disease evaluated and scored according to National Health Institute consensus staging | Up to 2 years
  The first day of chronic GVHD onset will be used to calculate the cumulative incidence. Calculated using the Gray method with prior death or relapse considered competing events.
Engraftment (recovery of granulopoiesis and megakaryopoiesis) | Up to 2 years
Incidence of infection | Up to day 100 post-transplant
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.
Non-relapse mortality defined as death occurring in a patient from causes other than relapse or progression | From date of stem cell infusion until non-disease related death, or last follow-up, whichever comes first, assessed up to 2 years
  The cumulative incidence of relapse/progression and non-relapse mortality will be calculated as competing risks using the Gray method. Descriptive statistics will also be used to assess the possible relationship between pre-HSCT disease status and outcomes. As the results of these evaluations are considered hypothesis-generating in nature, the statistics used will not include any formal statistical tests/comparisons.
Overall survival | Time from the day of stem cell infusion until death, or last follow-up, whichever comes first, assessed up to 2 years
  Estimate will be calculated using the Kaplan-Meier method.
Progression-free survival | date of stem cell infusion to the date of death, disease relapse/progression, or last follow-up, whichever occurs first, assessed up to 2 years
  Estimate will be calculated using the Kaplan-Meier method.
Relapse/progression | Up to 2 years
  The cumulative incidence of relapse/progression and non-relapse mortality will be calculated as competing risks using the Gray method. Descriptive statistics will also be used to assess the possible relationship between pre-hematopoietic stem cell transplant (HSCT) disease status and outcomes. As the results of these evaluations are considered hypothesis-generating in nature, the statistics used will not include any formal statistical tests/comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Haris Ali, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States